CLINICAL TRIAL: NCT02491775
Title: Genomic Landscape of EGFR Mutant NSCLC Prior to Afatinib and at the Time of Disease Progression Following Afatinib
Brief Title: Afatinib Genomic Landscape
Status: Terminated | Type: Observational
Why Stopped: Changes in treatment plan affecting drug therapy choices
Sponsor: Washington University School of Medicine (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 201408008
Record Dates: First submitted 2015-06-15; First posted 2015-07-08 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Non-small Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose to conduct a pilot feasibility study of single agent afatinib in patients with previously untreated metastatic EGFR (epidermal growth factor receptor) mutant adenocarcinoma of the lung (NSCLC = non-small cell lung cancer) with the sole purpose of characterizing the genomic landscape before afatinib and at the time of disease progression.

DETAILED DESCRIPTION:
The current proposal will include exome and transcriptome sequencing from blood collected at baseline along with tumor samples obtained prior to starting afatinib and at the time of disease progression (a total of two tissue samples and one blood sample per patient). The samples will be collected via consent to the IRB (Institutional Review Board) approved banking study "Tissue and Blood Acquisition for Genomic Analysis and Collection of Health Information from Patients with Thoracic Malignancies, Suspected Thoracic Malignancies, or Mesothelioma".

If carried out successfully, the proposed strategy very likely will lead to a larger and adequately powered study (perhaps using whole genome sequencing) to understand fully evolving molecular changes due to clonal selection under treatment pressure. The pace of progress in the field of sequencing technology currently underway is only likely to accelerate in the near future yielding richer and highly content-rich information. Moreover, it is likely that genomic information from DNA sequencing and transcriptome will be supplemented by analyses of translatomes and proteomes.

Successful completion of the proposed study would enable future studies to fully harness the potential of emerging technologies to develop novel approaches to treat and even ideally prevent resistance to EGFR TKIs (tyrosine-kinase inhibitor) and other molecularly targeted therapies. This could serve as a template for other cancer types as well. Over time, this approach, broadly used, would create simultaneously, highly valuable annotated tumor specimens along with germ line DNA for high-throughput genomic studies to identify novel targets and their impact on the course of disease. Re-analyzing molecular changes in the tumor at the time of disease progression would likely be a new standard of care to guide salvage therapy.

ELIGIBILITY:
Inclusion Criteria/Exclusion Criteria:

* Diagnosis of metastatic stage IIIB/IV lung adenocarcinoma
* Presence of known sensitizing mutations in EGFR TK domain (exon 19 deletion and L858R)
* Absence of known resistant mutations in the EGFR TK domain (T790M)
* Consented to HRPO # 201305031 ("Tissue and Blood Acquisition for Genomic Analysis and Collection of Health Information from Patients with Thoracic Malignancies, Suspected Thoracic Malignancies, or Mesothelioma")
* No prior treatment for this malignancy
* No prior localized therapy to the biopsy site
* Planned treatment with standard of care afatinib at 40 mg QD (daily)
* Not pregnant or breastfeeding
* At least 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the Washington University School of Medicine and Barnes-Jewish healthcare system who previously consented to study HRPO (Human Research Protection Office)# 201305031 ("Tissue and Blood Acquisition for Genomic Analysis and Collection of Health Information from Patients with Thoracic Malignancies, Suspected Thoracic Malignancies, or Mesothelioma").
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Genetic changes associated with disease progression following treatment with afatinib | Estimated to be 1 year
  * The investigators will compare tumor sequencing prior to afatinib treatment to the time of disease progression to see if the genetic sequencing changed between pre-treatment and progression.
  * The investigators plan to conduct exome and transcriptome sequencing of tumor before therapy with afatinib and at the time of relapse. In addition, exome sequencing of peripheral blood DNA will be done (for germline). Given the complexities of genomic analyses of paired samples in the face of limited data, the investigators will not be able to do any formal power calculations in this feasibility study.
  * Disease progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.

SECONDARY OUTCOMES:
Types of mutations in signaling kinases associated with therapeutic response | Estimated to be 1 year
  * Investigators will look at tumor tissue associated with a therapeutic response and compare with tumor tissue associated with disease progression and see if there are any mutation differences.
  * Therapeutic Response
    * Complete response is disappearance of all target lesions and non-target lesions.
    * Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Allelic ratio of wild type to mutant EGFR (roughly corrected for intrinsic differences in tumor cellularity) with duration of response | Estimated to be 1 year
  * A variant is considered to have mutant biased expression if the variant is expressed and the variant allele frequency is greater than 20% higher in the RNA-seq data compared to the exome sequencing data. A variant is considered to have wild type biased expression if the gene is expressed, the region of the variant is covered at 5X or greater depth, and the VAF is at least 20% lower in the RNA-seq data compared to the exome sequencing data.
  * Duration of response is the duration of overall response is measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu